CLINICAL TRIAL: NCT06142565
Title: Treatment of Postviral Olfactory Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Johan Lundström, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-03779-01; 2021-06527 (Other Grant/Funding Number: Swedish Research Foundation)
Record Dates: First submitted 2023-11-08; First posted 2023-11-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hyposmia
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Olfactory training with nose plugs (Experimental): Participants will complete olfactory training with scented nose plugs.
  Interventions: Device: Nose plug
- Olfactory training with household odors (Active Comparator): Participants will complete olfactory training with odors found in their household.
  Interventions: Other: Regular olfactory training

INTERVENTIONS:
Device: Nose plug — Participants will complete olfactory training with scented nose plugs.
  Arms: Olfactory training with nose plugs
Other: Regular olfactory training — Participants will complete olfactory training with regular odors found in their home.
  Arms: Olfactory training with household odors

SUMMARY:
A decreased sense of smell (hyposmia) is often caused by viral infections, such as COVID-19. Today, the only recommended treatment for hyposmia is olfactory training, a time consuming method with limitations in terms of both compliance and effect. The aim of this study is therefore to evaluate, as well as optimize, a new treatment method for olfactory loss.

Hyposmic participants will be recruited and randomized into two different treatment conditions. One group will do regular olfactory training and the other will do passive olfactory training with scented nose plugs. The training will be conducted in the home of the individual monday through friday for two consecutive months. Subjective and objectvie measures of olfactory problems will be assessed before and after treatment, as well as subjective measures related to quality of live and genereal wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years old
* Physically and cognitively capable of participating in the study
* Having appropriate olfactory screening test scores (hyposmic)

Exclusion Criteria:

* Anosmics
* Individuals with other diagnoses that could affect the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Objective olfactory function | 2 months
  Does the use of scented nose plugs increase the effect of olfactory training on objective olfactory function compared to regular olfactory training? For this outcome, we will use the standardized Sniffin' Sticks test to assess olfactory function.
Subjective symptoms and social/emotional consequences | 2 months
  Does the use of scented nose plugs increase the effect of olfactory training on subjective symptoms and social/emotional consequences compared to regular olfactory training? For this outcome, we will use the Sino-Nasal Outcome Test (SNOT).
Subjective health | 2 months
  Does the use of scented nose plugs increase the effect of olfactory training on subjective health compared to regular olfactory training? For this outcome, we will use the Self-Rated Health 5 measure and SF-36.
Subjective olfactory function | 2 months
  Does the use of scented nose plugs increase the effect of olfactory training on subjective olfactory function compared to regular olfactory training? For this outcome, we will use the Self-Reported Mini Olfactory Questionnaire.
Subjective degree of suffering from olfactory impairment | 2 months
  Does the use of scented nose plugs increase the effect of olfactory training on subjective degree of suffering from olfactory impairment compared to regular olfactory training? For this outcome, we will use the Questionnaire of Olfactory Disorders - Negative Statements.
Subjective parosmia | 2 months
  Does the use of scented nose plugs increase the effect of olfactory training on subjective parosmia compared to regular olfactory training? For this outcome, we will use the Landis parosmia questionnaire.
Subjective depressive symptoms | 2 months
  Does the use of scented nose plugs increase the effect of olfactory training on depressive symptoms compared to regular olfactory training? For this outcome, we will use the Beck Depression Inventory (BDI).
Subjective general wellbeing | 2 months
  Does the use of scented nose plugs increase the effect of olfactory training on depressive symptoms compared to regular olfactory training? For this outcome, we will use the General Well Being Schedule.
Compliance | 2 months
  Does the use of scented nose plugs increase the compliance of olfactory training compared to regular olfactory training? For this outcome, we will use questions asking the participants about their experience during the olfactory training, specifically targeting their compliance, such as how often they actually completed the olfactory training and how often they forgot to.

CONTACTS AND LOCATIONS:
Overall Officials: Johan N Lundstrom, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Winter AL, Henecke S, Thunell E, Swartz M, Martinsen J, Sahlstrand Johnson P, Lundstrom JN. Olfactory training using nasal inserts is more effective due to increased adherence. Rhinology. 2025 Aug 1;63(4):477-485. doi: 10.4193/Rhin24.369. PMID 40278843